CLINICAL TRIAL: NCT03007238
Title: Phase II Trial of Extracorporeal Photopheresis (ECP) Plus Low Dose IL-2 for Treatment of Steroid Refractory Chronic Graft-versus-Host Disease (cGVHD)
Brief Title: Extracorporeal Photopheresis and Low Dose Aldesleukin in Treating Patients With Steroid Refractory Chronic Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15125; NCI-2015-01933 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15125 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-11-23; First posted 2017-01-02 (Estimated); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — aldesleukin; Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (aldesleukin and ECP) (Experimental): Patients receive aldesleukin SC daily for 12 weeks. Patients also undergo ECP twice weekly on weeks 1-4 and then receive 2 ECP treatments every 2 weeks on weeks 5-12. Patients responding to upfront therapy with aldesleukin and ECP have the option to continue combination therapy per the discretion of the treating physician until clinical benefit is maintained or toxicities develop.
  Interventions: Biological: Aldesleukin; Procedure: Extracorporeal Photopheresis; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Procedure: Extracorporeal Photopheresis — Undergo ECP
  Other Names: Extracorporeal Photophoresis; photopheresis; Photophoresis
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies efficacy of extracorporeal photopheresis and low dose aldesleukin (interleukin-2) in treating patients with chronic graft-versus-host disease (cGVHD) that does not respond to upfront treatment with steroids. In graft-vs-host disease, patients have a small quantity of a white blood cell called T regulatory cells or T-reg cells that helps to control the immune system. Extracorporeal photopheresis is a procedure where patient's blood is removed and treated with ultraviolet light and drugs that become active when exposed to light. The treated blood is then returned to the patient and may be effective in increasing T-reg cells in patients with cGVHD. Aldesleukin increases the activity and growth of white blood cells, and it has shown to enhance T-reg cells in patients with cGVHD and may be effective improving GVHD symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the anti-cGVHD activity of extracorporeal photopheresis (ECP) when combined with low dose IL-2 (interleukin 2) (aldesleukin), in patients with steroid refractory cGVHD, as assessed by overall cGVHD response rate (complete response [CR]+partial response [PR]+stable disease [SD]).

SECONDARY OBJECTIVES:

I. Characterize and evaluate toxicities, including type, frequency, severity, attribution, time course and duration.

II. Estimate overall and failure-free survival, non-relapse mortality (NRM) and relapse, through 1 year after initiation of treatment.

III. Characterize chronic GVHD Symptom Scale scores -self-report (with assistance from register nurses [RNs] and medical doctors [MDs]).

IV. Assess the immunologic effects of low-dose daily subcutaneous (SC) IL-2 + ECP.

V. Correlate clinical endpoints of response with ECP performance parameters.

OUTLINE:

Patients receive aldesleukin subcutaneously (SC) daily for 12 weeks. Patients also undergo ECP twice weekly on weeks 1-4 and then receive 2 ECP treatments every 2 weeks on weeks 5-12. Patients responding to upfront therapy with aldesleukin and ECP have the option to continue combination therapy per the discretion of the treating physician until clinical benefit is maintained or toxicities develop.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of allogeneic stem cell transplantation with myeloablative or non-myeloablative conditioning regimens; alternative donor transplants (umbilical cord blood and haploidentical) are allowed
* Patients with chronic GVHD requiring systemic therapy are eligible
* Participants must have steroid-refractory cGVHD, which is defined as having persistent signs and symptoms of cGVHD despite the use of prednisone at 0.20 mg/kg/day (or 0.5 mg/kg every other day) for at least 4 weeks (or equivalent dosing of alternate corticosteroids) without complete resolution of signs and symptoms
* Karnofsky performance status of 70-100 %
* Estimated life expectancy greater than 3 months
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Stable dose of corticosteroids for 2 weeks prior to enrollment, i.e. the patient's steroid dose (mg/kg) will remain unchanged (eg 0.5 mg/kg) in the 2 weeks preceding enrollment; allowances will be made for up or down titrating the dose based on changes in body weight
* Total bilirubin < 2.0 mg/dl-exception permitted in patients with Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x upper limit of normal (ULN), unless hepatic dysfunction is a manifestation of presumed cGVHD
* Abnormal liver function tests (LFTs) in the context of active cGVHD involving other organ systems may also be permitted if the treating physician documents the LFTs as being consistent with hepatic cGVHD and a liver biopsy will not be mandated in this situation
* Serum creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal
* Absolute neutrophil count (ANC) > 1000/mm^3
* Platelets > 50,000/mm^3
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Patients with steroid refractory cGVHD typically have received salvage with multiple lines of therapy; hence in this trial there will be no restriction in terms of prior lines of therapy received; prior ECP exposure is allowed, however prior IL-2 use is excluded

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection; patients with an ongoing prednisone requirement of > 1 mg/kg/day (or equivalent) will be excluded
* History of thrombotic microangiopathy, hemolytic-uremic syndrome or thrombotic thrombocytopenic purpura
* Exposure to any new immunosuppressive medication in the 4 weeks prior to enrollment
* Donor lymphocyte infusion within 100 days prior to enrollment
* Active malignant relapse
* Uncontrolled cardiac angina or symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV)
* Human immunodeficiency virus (HIV)-positive individuals on combination antiretroviral therapy are ineligible
* Patients may not be receiving any other investigational agents, or concurrent parenteral biological, chemotherapy, or radiation therapy. Oral chemotherapeutic agents or biologics-for example ruxolitinib therapy (either past or current exposure)-is allowed
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to IL-2
* Patients must not have received prior chemotherapy (pentostatin) within 4 weeks before study enrollment, and those who have not recovered from the adverse events due to agents administered more than 4 weeks earlier are excluded
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with IL-2
* Patients with other active malignancies are ineligible for this study, other than superficial localized skin cancer (basal or squamous cell carcinoma)
* Subjects, who in the opinion of the investigator may not be able to comply with IL-2 or ECP treatment requirements or the safety monitoring requirements of the study, will be excluded from participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Salhotra, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Patients received ECP twice weekly for weeks 1 through 4, then two treatment every other week until week 12 of protocol therapy. Daily IL-2 was given subcutaneously for 12 weeks. GVHD assessments were done at the baseline, then at 3-weeks intervals at 3, 6, 9,12 and 16 weeks.
Period: Overall Study
Arm/Group | Overall Study
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 10 participants
Groups:
- Treatment (ECP Plus Low Dose IL-2): Patients also undergo ECP twice weekly on weeks 1-4 and then receive 2 ECP treatments every other week until week 12 of protocol therapy. Patients receive aldesleukin subcutaneously (SC) daily for 12 weeks.
  Patients responding to upfront therapy with aldesleukin and ECP have the option to continue combination therapy per the discretion of the treating physician until clinical benefit is maintained or toxicities develop.
  After completion of study treatment, patients are followed up periodically.
Arm/Group | Treatment (ECP Plus Low Dose IL-2)
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 46 [22 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate at Week 16 (4 Weeks After the End of Treatment)
Description: Defined as the proportion of response-evaluable participates that achieve a CR/PR or SD at Week 16 (4 weeks after the end of treatment).
Time Frame: At Week 16 (4 weeks after the end of treatment)
Population: At week 16, nine of the ten patients were alive and evaluable for response assessment. ORR was calculated for nine patients who were alive at Week 16 and was also calculated by ITT for ten patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (ECP+IL-2): Patients received ECP twice weekly for weeks 1 through 4, then two treatment every other week until week 12 of protocol therapy. Daily IL-2 was given subcutaneously for 12 weeks. GVHD assessments were done at the baseline, then at 3-weeks intervals at 3, 6, 9,12 and 16 weeks.
Arm/Group | Treatment (ECP+IL-2)
Number analyzed (Participants) | 10
percentage of participants
  Overall response rate in patients who were alive at Week 16 (4 weeks after the end of treatment): number analyzed (Participants) | 9
  Overall response rate in patients who were alive at Week 16 (4 weeks after the end of treatment) | 88.9 [51.8 to 99.7]
  Overall response rate by ITT | 80.0 [44.4 to 97.5]

2. Secondary Outcome: Failure-free Survival
Description: Failure-free survival will be estimated using the product-limit method of Kaplan and Meier.
Time Frame: From date of first dose of study drug to first documented cGVHD progression (necessitating change of treatment), malignancy relapse or progression or death from any cause, whichever occurs first, assessed up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Overall Study: Patients received ECP twice weekly for weeks 1 through 4, then two treatment every other week until week 12 of protocol therapy. Daily IL-2 was given subcutaneously for 12 weeks. Patients' survival was follow through 1 year after initiation of treatment.
Arm/Group | Overall Study
Number analyzed (Participants) | 10
percentage of participants | 40 [18.7 to 85.5]

3. Secondary Outcome: Overall Survival
Description: Overall survival was estimated using the product-limit method of Kaplan and Meier.
Time Frame: From date of first dose of study drug to date of death from any cause, assessed up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 10
percentage of participants | 60 [36.2 to 99.5]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from date of first dose of study drug up to 16 weeks. All-Cause Mortality was assessed from first dose until death, assessed up to 1 year.
Groups:
- Overall Study: To evaluate the anti-cGVHD activity of extracorporeal photopheresis (ECP) when combined with low dose IL-2 (interleukin 2) (aldesleukin), in patients with steroid refractory cGVHD, as assessed by overall cGVHD response rate (complete response [CR]+partial response [PR]+stable disease [SD]).
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 4/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=10)
Atrial flutter (Cardiac disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=10)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Anal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03007238/Prot_SAP_000.pdf